CLINICAL TRIAL: NCT04444973
Title: Use of Right Ventricular Conductance Catheter Guidance to Optimise Balloon Pulmonary Angioplasty as a Non Surgical Treatment of Chronic Thromboembolic Pulmonary Hypertension.
Brief Title: RV Conductance Catheter Assessment During Balloon Pulmonary Angioplasty
Acronym: RVBPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 229599
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Balloon pulmonary angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive RV assessment: RV conductance catheter assessment of RV performance
  Interventions: Procedure: Balloon pulmonary angioplasty

INTERVENTIONS:
Procedure: Balloon pulmonary angioplasty — Balloon dilatation of sub segmental pulmonary artery web disease

SUMMARY:
Balloon pulmonary angioplasty (BPA) treats patients with inoperable chronic thromboembolic pulmonary hypertension (CTEPH). Intra-procedural markers of success to guide the intervention are lacking. The investigators propose to measure right ventricular (RV) pressure volume loops invasively and measure biomarkers at intervals during the course of a course of BPA. These data will be analysed to define load independent indices of RV functional improvement, cross correlated with biomarker data and be used to calibrate non-invasive assessment of ventriculo-arterial coupling by cardiac magnetic resonance imaging (CMR) to better detect responders of BPA and pulmonary endarterectomy (PEA).

DETAILED DESCRIPTION:
Patients who have Chronic Thromboembolic Pulmonary Hypertension (CTEPH) can treated surgically or by undergoing minimally invasive balloon pulmonary angioplasty (BPA). However not all patients have resolution of their pulmonary hypertension following these procedures, and some patients who don't have pulmonary hypertension derive substantial benefit nonetheless from surgical clearance of their thromboembolic disease.

Thus better understanding of the interaction between the blood vessels, the right heart workload, and symptoms and outcomes is required to predict treatment response. Ventriculo-arterial coupling is one such measure, quantifying the efficiency of transfer of energy from the right ventricle to the pulmonary arteries. Traditionally this has required invasive procedures involving intracavity conduction catheterisation of the right ventricle to simultaneously measure flow and pressure whilst altering preload. Not only is this invasive, but it is not routinely performed in clinical practice due to its complexity and requirement for specialised expertise and equipment. As CMR can simultaneously assess right ventricular and pulmonary function it may be able to assess function and ventriculo-arterial coupling non-invasively and allow for a more detailed and accessible mode of disease quantification and stratification.

The investigators will measure how the right heart function changes during BPA in patients with inoperable CTEPH, measured using a conductance catheter placed within the pumping chamber on the right side of the heart (right ventricle). This will generate pressure volume loops to detect intra-procedural changes of ventriculo-arterial coupling that can be used to quantify treatment success. The investigators will also monitor the levels of a newly discovered vessel inflammatory marker in the blood - Angiopoietin 2 (Ang2), and N-terminal pro-brain natriuretic peptide (NT-Pro BNP) that may also be useful in identifying responders to treatment and help define the optimal treatment protocol for BPA.

This participants will have CMR as standard of care. Data from CMR and invasive measurements of ventriculo-arterial coupling will determine the best CMR measures of coupling efficiency. These measures will then be applied within a large well-characterised cohort with long term follow-up to determine its association with symptoms, and outcomes following surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Able to provide informed consent
* Inoperable CTEPH eligible for BPA treatment

Exclusion Criteria:

* Severe co-morbidity (expected life <6months)
* Women of child bearing age
* Significant known left to right shunt
* Permanent pacemaker
* Atrial fibrillation
* Severe lung parenchyma disease ( eg emphysema, Interstitial Lung Disease (ILD)).
* Retained metallic foreign body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable CTEPH undergoing BPA
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in RV Tau | 3 months
  Does BPA result in a significant change in right ventricular time constant of diastolic relaxation - a measure of diastolic dysfunction

SECONDARY OUTCOMES:
Ang2 an pro-NT BNP | 3 months
  Does Ang2 and pro-NT BNP correlate with invasively acquired pressure volume loop data
CMR | 3 months
  Does non-invasive ventriculo-arterial (VA) coupling by cardiac magnetic resonance imaging correlate with invasively derived pressure volume loop data

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Hoole, MD, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared